CLINICAL TRIAL: NCT07110545
Title: Effect of Acupuncture on Postoperative Pain Relief in Patients Undergoing Laparoscopic Cholecystectomy in Suez Canal University Hospitals: A Randomized Controlled Trial
Brief Title: Acupuncture on Postoperative Pain Relief in Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, professor of anaesthesia, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: acupunture in cholecystectomy
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Acupuncture; Postoperative Pain Management; Cholecystectomy, Laparoscopic
Keywords: acupuncture; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Active Comparator): Interventional group: included 25 patients for Acupuncture
  Interventions: Other: Acupuncture
- Control (No Intervention): Control patients: included 25 patients who received no intervention.

INTERVENTIONS:
Other: Acupuncture — Application of acupuncture on specific acupoints
  Arms: Acupuncture

SUMMARY:
To lessen related side effects, opioids are used as needed to treat pain after laparoscopic cholecystectomy (LC). Research into the efficacy of acupuncture as an adjunct treatment for postoperative patients has gained traction. However, the findings of these studies are inconsistent. It has been suggested that acupuncture may not influence postoperative pain, whereas studies involving various surgical procedures have reported favorable results. Nonetheless, there is scant evidence demonstrating the effectiveness of acupuncture in managing pain following LC. In order to assess the effectiveness and safety of acupuncture in reducing postoperative pain in patients following LC, this study was created.

The study's objective was to reduce postoperative pain in order to improve the results of LC surgeries.

Fifty patients participated in this prospective randomized controlled interventional study, split equally between two groups.

DETAILED DESCRIPTION:
One common minimally invasive surgical technique is laparoscopy, where minimizing postoperative pain and nausea and vomiting is of utmost importance. It necessitates early patient mobilization and short-term discharge due to its outpatient characteristics. With over 80% of surgical patients experiencing postoperative pain of varying intensities, postoperative pain presents a significant challenge for clinicians. One of the main reasons why hospital stays are prolonged is postoperative pain.

A number of pharmacological and nonpharmacological approaches, including transversus abdominis plane block, low-pressure pneumoperitoneum, and local anesthetics, have been clinically investigated to treat pain following LC; these approaches require additional research. Effective analgesics that are frequently used in the postoperative surgical phase are nonsteroidal anti-inflammatory drugs (NSAIDs). The use of NSAIDs may be restricted due to the associated risks of gastrointestinal harm and possible postoperative complications, such as bleeding, anastomotic leaks, and soft tissue infection.

Opioids are used as needed to treat pain following LC in order to prevent associated side effects.

Research on acupuncture's effectiveness as a postoperative adjuvant treatment has grown in popularity. The studies' findings, however, are not entirely consistent. Although studies using various surgical procedures produced positive results, it was suggested that acupuncture has no effect on postoperative pain. However, there is scant evidence regarding acupuncture's ability to manage pain following LC. Therefore, the purpose of this study was to investigate the safety and effectiveness of acupuncture in treating postoperative pain in patients following LC. Therefore, the study's goal was to reduce postoperative pain in order to enhance the results of LC surgeries.

Fifty patients, equally split into two groups, participated in this prospective randomized controlled interventional study.

* There were 25 patients in Group I (Interventional group) who received acupuncture.
* 25 patients in Group II (control patients) did not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing laparoscopic cholecystectomy of both sexes.
* Patients with grades I and II from the American Society of Anesthesiologists (ASA).

Exclusion Criteria:

* Patients with local skin infections at acupoints.
* Patients who have nerve injuries on upper limbs or lower limbs.
* Patients who are alcoholics.
* Pregnant.
* Patients with other severe systemic diseases and serious mental illnesses.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pethidine | From the moment the surgery was completed until 24 hours after the procedure
  The total amount of pethidine required to manage pain following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No